CLINICAL TRIAL: NCT03805763
Title: Clinical Research on the Effect of Different Extents of Internal Limiting Membrane Peeling on Macular Hole Closure and Visual Acuity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Xiangtian Zhou, Professor, Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZZD-Macular Hole
Record Dates: First submitted 2019-01-13; First posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Macular Holes
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Large extent of ILM Peeling (Experimental): Extent of ILM peeling is 4DD and the ILM flap is inserted
  Interventions: Procedure: Large extent of ILM Peeling
- Small extent of ILM Peeling (Experimental): Extent of ILM peeling is 2DD and the ILM flap is inserted
  Interventions: Procedure: Small extent of ILM Peeling

INTERVENTIONS:
Procedure: Large extent of ILM Peeling — The extent of ILM peeling is 4DD
  Arms: Large extent of ILM Peeling
Procedure: Small extent of ILM Peeling — The extent of ILM peeling is 2DD
  Arms: Small extent of ILM Peeling

SUMMARY:
Observing and describing the surgical effects of different extents of internal limiting membrane peeling combined with internal limiting membrane insertion for macular hole

ELIGIBILITY:
Inclusion Criteria:

* Clear diagnosis of macular hole;
* The minimum diameter of the macular hole is >400 μm;
* Without serious systemic disease that make patients can not be operated;

Exclusion Criteria:

* suffering from severe retinal diseases such as: diabetic retinopathy, age-related macular degeneration, peripheral retinal detachment, PVR, etc.;
* opacitas in the refractive medium can not perform Angio-OCT and visual acuity examination;
* eye acute and chronic inflammation, such as acute contagious conjunctivitis, acute and chronic keratitis, acute dacryocystitis;
* traumatic macular hole, secondary macular hole, high myopia macular hole, etc.;
* having a history of vitrectomy surgery;
* glaucoma in stage of preclinical, severe stenosis or closure;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Condition of postoperative healing of macular holes | 1 year
  postoperative photograph of macular retina scanned by Angiography Optical Coherence Tomography(AngioOCT)
Mean change from baseline in best-corrected visual acuity (BCVA) | 1 year
  Assessed using the ETDRS protocol
change from baseline in foveal avascular zone (FAZ) areas and diameter | 1 year
  Assessed on AngioOCT
change from baseline in the area and diameter of deteriorated circulation zone in superficial and deep retina vessels | 1 year
  Assessed on AngioOCT

CONTACTS AND LOCATIONS:
Overall Officials: Zongduan Zhang, M.D,PhD, Principal Investigator — The Eye Hospital of Wenzhou Medical University